CLINICAL TRIAL: NCT01311791
Title: A Randomized, Controlled Study to Evaluate the Safety and Cardiovascular Effects of Algisyl-LVR™ as a Method of Left Ventricular Augmentation in Patients With Dilated Cardiomyopathy (AUGMENT-HF)
Brief Title: A Randomized, Controlled Study to Evaluate Algisyl-LVR™ as a Method of Left Ventricular Augmentation for Heart Failure
Acronym: AUGMENT-HF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: LoneStar Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LSH-10-001
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure; Dilated Cardiomyopathy
Keywords: Left ventricular augmentation; Left ventricular restoration
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Algisyl-LVR (Experimental): Algisyl-LVR™ device (implants) administered during a surgical procedure.
  Interventions: Device: Algisyl-LVR
- Standard Medical Therapy (Active Comparator): as per protocol
  Interventions: Drug: Standard medical therapy

INTERVENTIONS:
Device: Algisyl-LVR — Algisyl-LVR™ device (implants) administered during a surgical procedure
  Other Names: intramyocardial injections of Alginate hydrogel
  Arms: Algisyl-LVR
Drug: Standard medical therapy — as defined per protocol
  Other Names: evidence-based therapy for heart failure; heart failure medications; drug therapy
  Arms: Standard Medical Therapy

SUMMARY:
This is a pilot study to evaluate the safety and efficacy of the Algisyl-LVR™ device. The purpose of this study is to investigate Algisyl-LVR™ employed as a method of left ventricular augmentation and restoration in patients with dilated cardiomyopathy. Algisyl-LVR™ will be injected into the myocardium under direct visualization during the surgical procedure.

This study will evaluate the concept that direct mid left ventricular (LV) intramyocardial injections of Alginate hydrogel implants into the free wall of the failing LV will reduce LV size, restore LV shape, lower LV wall stress and improve global LV function.

The Primary Efficacy Endpoint of the study is the change in Peak VO2 (maximum oxygen uptake) from baseline to 6 months of follow-up. The Primary Safety Endpoint of the study is to estimate the 30 day mortality associated with the implantation of the Algisyl-LVR device

The hypothesis of the study is that there is a statistically significant difference in change in Peak VO2 from baseline to 6 month follow-up when the medically managed arm is compared to the Algisyl-LVR arm, i.e. the Algisyl LVR arm is superior to medical management.

DETAILED DESCRIPTION:
This is a prospective, randomized, parallel group evaluation of the safety and effectiveness of Algisyl-LVR in patients with dilated cardiomyopathy of either ischemic or non-ischemic origin. The evaluation for primary efficacy endpoint (Peak VO2) at 6 months will be investigator-blinded. The primary safety endpoint, while not blinded, is 30 day all-cause mortality and an objective assessment. The remaining study endpoints will evaluate the effects of the device through the evaluation of functional, structural, biochemical, and electrocardiographic evaluations at 6 and 12 months. Evaluation of adverse events and these assessments will also provide evidence of the safety profile of the device in patients with dilated cardiomyopathy.

Pre-enrollment baseline patient evaluation will include clinical assessment, assessment of New York Heart Association (NYHA) functional class, blood tests, chest x-ray, echocardiography, magnetic resonance imaging (MRI), electrocardiogram, cardiopulmonary exercise testing, submaximal exercise testing, and quality of life assessments. Blinded central evaluation will be performed for measures of cardiopulmonary exercise testing, blood tests, Holter Monitors and cardiac imaging.

After written patient informed consent has been obtained and verification of eligibility, patients who meet the selection criteria will be randomized. All patients must be on stable, evidence-based therapy for heart failure. Patients assigned to the Investigational Device group will have the Algisyl-LVR™ device (implants) administered during a surgical procedure. For patients randomized to the investigational device group, the investigator will make every attempt to minimize the time between randomization and surgery (i.e, no more than 7 to 10 days). Patients will be considered part of the study cohort as soon as they have been randomly allocated to either the Treatment or Control group. This time point will also be considered as the start of follow-up. For patients allocated to the Investigational Device group, the starting point of follow-up for surgical mortality and surgical complications will start as of the date when the surgical procedure is performed (or attempted). The acute response to device implant will be monitored intraoperatively via continuous electrocardiographic cardiac monitoring, arterial pressure lines, transesophageal echocardiography (TEE), and pulmonary artery catheter. Patients receiving the investigational device are expected to remain hospitalized for 5 to 14 days. Patients assigned to the control group will continue on standard medical therapy (without the investigational device).

Follow-up in this study is divided into two phases. During the first phase, referred to as the "efficacy phase", repeat testing of patient functional and cardiac structural parameters will be conducted at follow-up visits scheduled at 3 months and 6 months, and every 6 months thereafter. Follow-up testing will be supplemented by a 30 day (post randomization) telephone contact with all patients. The efficacy phase of the trial will end on a common closing date after a minimum of 6 months of follow-up (i.e., after the last patient enrolled has been completed the 6 month visit). At that point data analysis will be performed and an initial study report will be generated. Following completion of the efficacy phase, long-term monitoring will continue through each patient's 24-month visit. This second phase is referred to as the "extended follow-up phase". During this phase, data collection will be focused on long-term safety and will be conducted at 6-month intervals.

Patient's randomized to the control group and completing the 12 month visit will be provided the option of enrolling in Clinical Study LSH-11-001: An Open Label Rollover Trial for Patients Randomized to the Control Group of Study LSH-10-001. Patients must continue to meet the inclusion and exclusion criteria as stated in Study LSH-10-001 to be eligible for Study LSH-11-001.

ELIGIBILITY:
Inclusion Criteria:

1. The patients must be able and willing to give written informed consent
2. The patients will be adult (age ≥ 18 years and ≤ 79 years) males or females
3. The patients must be on stable, evidence-based therapy for heart failure

   * Note: CRT or CRT-D are acceptable co-therapy, if placed > 3 months before randomization or the investigator does not anticipate within 6 months after randomization
4. The patients will have a left ventricular ejection fraction equal to or less than 35% via echocardiography, cardiac catheterization, radionuclide scan, or magnetic resonance imaging (measured within the last 30 days)
5. The patients will have a left ventricular end diastolic dimension indexed to body surface area (LVEDDi) of 30 to 40mm/m2 (LVEDD/BSA) (measured within the last 30 days)
6. Patients must have symptomatic heart failure with a Peak VO2 of 9.0 - 14.5 ml/min/kg (performed using a bicycle ergometer). Patients must perform two CPX tests (within 30 days of randomization and performed at least 20 hours apart) that differ by no more than 15% in the observed value for Peak VO2 and have a mean value of 9.0 - 14.5 ml/min/kg from these two tests.
7. Patient's surgical risk must be considered reasonable and the evaluation of surgical risk should include review of coronary and left ventricular angiography
8. If female, the patients must be (a) post-menopausal, (b) surgically sterile, or (c) using adequate birth control and have a negative serum pregnancy test within 7 days prior to administration of study device

Exclusion Criteria:

1. Patients for whom it is planned to receive CABG, MVR, heart transplantation or LVAD within the next 6 months.
2. Patients presenting with cardiogenic shock.
3. Patients who have undergone a previous mid-sternotomy surgical procedure are excluded unless the surgeon's assessment is that the left sided limited thoracotomy is feasible and considered reasonable surgical risk.
4. Patients presenting with a restrictive cardiomyopathy such as due to amyloidosis, sarcoidosis, or hemochromatosis
5. Patient with a history of constrictive pericarditis
6. Patients with a Q wave myocardial infarction (MI) within the last 30 days
7. Patients with a recent history of stroke (within 60 days prior to the surgical procedure)
8. A left ventricular (LV) wall thickness of the LV free-wall, at the mid-ventricular level, of less than 8 mm (screening echocardiography must confirm a minimum wall thickness of 8 mm)
9. Patients with a serum creatinine > 2.5 mg/dL
10. Clinically significant liver enzyme abnormalities, i.e., AST(SGOT) and ALT (SGPT) more than 2.5 times the upper limit of normal
11. History of severe COPD (i.e., FEV 1< 1 liter or FEV1 < 50% predicted)
12. The patients will not be receiving concurrently an investigational Product in another clinical trial or have received an investigational Product in another clinical trial in the 30 days prior to enrollment
13. A life expectancy of less than 1 year or any other condition that, in the opinion of the clinical investigator, might compromise any aspect of the trial

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
peak VO2 | 6 months
  The primary effectiveness endpoint will be a comparison of change in Peak VO2 from baseline to 6 months of follow-up between the Algisyl-LVR and medically managed arms with the intention to prove superiority in improvement in Peak VO2 associated with the Algisyl-LVR study group as compared to the medically managed study group. Evaluation of the cardiopulmonary exercise testing will be conducted by a central, blinded core laboratory.

SECONDARY OUTCOMES:
30 day all cause mortality | 30 days
  The primary safety objective is to estimate the 30 day cardiac mortality associated with the implantation of the Algisyl-LVR device and qualitatively compare the observed rate to literature estimates for similar patients undergoing cardiac surgeries comparable in risk to implantation of the Algisyl-LVR

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Volterani, MD, Principal Investigator — IRCCS San Raffaele Pisana
Locations (18):
- Heart Center at the Alfred, Melbourne, Victoria, Australia
- Germany (5):
  - Charité (Campus Virchov), Berlin
  - Charité - Universitätsmedizin Berlin (Campus Benjamin Franklin), Berlin
  - Herzzentrum Dresden Universitätsklinik, Dresden
  - Universität Schleswig-Holstein Campus Kiel, Kiel
  - Universitätsklinikum Ulm, Ulm
- Italy (7):
  - IRCCS Policlinico San Donato, San Donato, Milanese (MI)
  - IRCCS San Raffaele Roma, Rome, Rome
  - Ospedali riuniti Dipartimento Cardiovascolare, Bergamo
  - Istituti Ospitalieri di Cremona, Cremona
  - Istituto Scientifico Universitario San Raffaele, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Policlinico Umberto I, Rome
- St. Antonius Ziekenhuis Nieuwegein, Nieuwegein, Netherlands
- Auckland City Hospital, Auckland, New Zealand
- Romania (3):
  - Centrului Clinic de Urgenta de Boli Cardiovasculare al Armatei, Bucharest
  - Clinica de Cardiologie, Spitalul Clinic de Urgenta "Sf. Pantelimon", Bucharest
  - Spitalul Clinic De Urgenta MAI "Prof. Dr. Dimitrie Gerota", Bucharest

REFERENCES:
- [Result] Anker SD, Coats AJ, Cristian G, Dragomir D, Pusineri E, Piredda M, Bettari L, Dowling R, Volterrani M, Kirwan BA, Filippatos G, Mas JL, Danchin N, Solomon SD, Lee RJ, Ahmann F, Hinson A, Sabbah HN, Mann DL. A prospective comparison of alginate-hydrogel with standard medical therapy to determine impact on functional capacity and clinical outcomes in patients with advanced heart failure (AUGMENT-HF trial). Eur Heart J. 2015 Sep 7;36(34):2297-309. doi: 10.1093/eurheartj/ehv259. Epub 2015 Jun 16. PMID 26082085
- [Result] Mann DL, Lee RJ, Coats AJ, Neagoe G, Dragomir D, Pusineri E, Piredda M, Bettari L, Kirwan BA, Dowling R, Volterrani M, Solomon SD, Sabbah HN, Hinson A, Anker SD. One-year follow-up results from AUGMENT-HF: a multicentre randomized controlled clinical trial of the efficacy of left ventricular augmentation with Algisyl in the treatment of heart failure. Eur J Heart Fail. 2016 Mar;18(3):314-25. doi: 10.1002/ejhf.449. Epub 2015 Nov 11. PMID 26555602